CLINICAL TRIAL: NCT01929837
Title: Treatment of Tinnitus With Transcranial Magnetic Stimulation
Brief Title: Tinnitus rTMS 2013
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: Satakunta Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: T69/2013
Record Dates: First submitted 2013-06-24; First posted 2013-08-28 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Tinnitus
Keywords: Tinnitus; Transcranial magnetic stimulation
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- E-fied navigated rTMS (Experimental): Electrical field navigated transcranial magnetic stimulation
  Interventions: Device: E-fied navigated rTMS
- sham E-field navigated rTMS (Sham Comparator): Sham electrical field navigated rTMS
  Interventions: Device: sham E-field navigated rTMS
- non-navigated rTMS (Experimental): non-navigated rTMS
  Interventions: Device: non-navigated rTMS
- Experimental, Navigated rTMS (Experimental): Navigated rTMS,
  Interventions: Device: Navigated rTMS

INTERVENTIONS:
Device: E-fied navigated rTMS — 1 hz on the superior temporal gyrus contralateral/left side with E-field navigated rTMS (Nexstim) targeted at the tonotopic representation area of the main frequency content of tinnitus
  Arms: E-fied navigated rTMS
Device: non-navigated rTMS — 1 hz on the superior temporal gyrus contralateral/left side with non-navigated rTMS according to external landmarks (between T3/T4 and P3/P4 EEG-electrode locations)
  Arms: non-navigated rTMS
Device: sham E-field navigated rTMS
  Arms: sham E-field navigated rTMS
Device: Navigated rTMS — 1 hz on the left superior temporal gyrus with (MRI) navigated rTMS (Visor)
  Arms: Experimental, Navigated rTMS

SUMMARY:
Tinnitus is the perception of sound in the absence of corresponding external sound. Tinnitus affects approximately 10-15 % of the population. The prevalence increases with age and it is estimated that more than 20 % of the older people have tinnitus. Approximately 10-15 % of tinnitus patients have clinically relevant, disabling tinnitus causing for example anxiety, depression and sleep disturbances. The treatment of chronic tinnitus is difficult and most therapies focus on alleviating the condition rather than treating the cause. Pathophysiology of tinnitus still remains incompletely understood. Functional brain imaging data in tinnitus patients and animal models suggest that tinnitus is associated with increased neuronal activity, increased synchronicity, and functional reorganization within the auditory cortex either uni- or bilaterally, but there are also functional alterations in brain areas outside the auditory system. Transcranial magnetic stimulation (TMS) is a neuromodulation technique based on the principle of electromagnetic induction of an electric field in the brain by means of magnetic pulses given to the scalp. TMS is a non-invasive, painless, and safe method for modulation of cortical activity. TMS pulses given at low frequencies (≤ 1 Hz) have been shown to decrease cortical excitability both in experimental settings and humans, which forms the basis for using low frequency rTMS to treat chronic tinnitus patients, in whom hyperactivity of the auditory cortex has been observed in functional brain imaging studies

ELIGIBILITY:
Inclusion Criteria:

* chronic tinnitus 6 months-10 years
* age 18-65 years
* tinnitus intensity VAS at least 4/10

Exclusion Criteria:

* pulsatile tinnitus
* objective tinnitus
* epilepsy, brain disease
* severe/recent heart disease
* pregnancy
* alcohol abuse
* metallic implants etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-09; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
The change of loudness and pitch of the tinnitus is psychophysically measured, VAS questionnaires, Tinnitus Handicap Inventory, Tinnitus diary | Change from baseline and 2-3 days after treatment period

CONTACTS AND LOCATIONS:
Locations (1):
- Turku University Hospital, Turku, Southwest Finland, Finland

REFERENCES:
- [Derived] Sahlsten H, Taiminen T, Karukivi M, Sjosten N, Nikkila J, Virtanen J, Paavola J, Joutsa J, Niinivirta-Joutsa K, Takala M, Holm A, Rauhala E, Loyttyniemi E, Johansson R, Jaaskelainen SK. Psychiatric (Axis I) and personality (Axis II) disorders and subjective psychiatric symptoms in chronic tinnitus. Int J Audiol. 2018 Apr;57(4):302-312. doi: 10.1080/14992027.2017.1409440. Epub 2017 Nov 30. PMID 29188734